CLINICAL TRIAL: NCT03408132
Title: A Phase Ib/IIa Open-label, Repeated Dose, Metabolic Balance Study of FE 203799 in Patients With Short Bowel Syndrome and Intestinal Insufficiency
Brief Title: Metabolic Balance Study of FE203799 in Patients With SBS With Intestinal Insufficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlyPharma Therapeutics (Industry)
Collaborators: VectivBio AG (Industry)
Responsible Party: Sponsor
Organization: VectivBio AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLY-321-2017
Record Dates: First submitted 2017-11-21; First posted 2018-01-23 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2020-02

CONDITIONS: SBS - Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FE203799 5 mg (Experimental): FE203799 5 mg subcutaneous injection
  Interventions: Drug: FE203799

INTERVENTIONS:
Drug: FE203799 — FE203799 5 mg subcutaneous once weekly
  Other Names: GLP 2 analogue

SUMMARY:
This is a repeated dose, open label trial investigating safety, efficacy, PD and PK of FE 203799 in 8 patients with SBS. The patients will receive a subcutaneous (SC) dose of 5 mg FE 203799 once weekly for 4 consecutive weeks, and efficacy parameters and PK will be assessed after the fourth dose. Safety follow up assessments will be performed 4-6 weeks after the last dose.

DETAILED DESCRIPTION:
This is a repeated dose, open label trial investigating safety, efficacy, PD and PK of FE 203799 in 8 patients with SBS . The patients will receive a subcutaneous (SC) dose of 5 mg FE 203799 once weekly for 4 consecutive weeks, and efficacy parameters and PK will be assessed after the fourth dose. Safety follow-up assessments will be performed 4-6 weeks after the last dose.

The first two administrations of trial drug will be performed at the clinic, while the third dose can be either self-administered by the patient or administered at the clinic if the patient prefers to travel to the site or other considerations make a site visit preferable. The fourth administration of trial drug will be performed at the clinic just prior to assessment of efficacy parameters in the treatment balance study.

Prior to each administration of trial drug, liver function parameters will be analysed and assessed. During the entire trial, patients who develop extremely high or persistently elevated liver enzymes following trial drug administration will be discontinued from the trial.

The patients will complete a diary with data on trial drug administration performed at home, local tolerability and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with SBS secondary to surgical resection of the small intestine, with or without an intact colon.
2. 18-80 years of age
3. Average faecal wet weight excretion of ≥1500 g/day during the baseline balance study
4. Average urine production <2000 mL/day during the baseline balance study
5. Body Mass Index (BMI) between 16.0 and 32.0 (both inclusive)
6. At least 6 months since last surgical bowel resection
7. Willing to adhere to a defined oral intake of fluids on certain days as required by the protocol (and based on the individual's routine daily consumption)
8. Women of childbearing potential must agree to use an adequate method of contraception during the trial and for 60 days after the end-of-trial visit. Adequate methods of contraception include intrauterine device or hormonal contraception (oral contraceptive pill, depot injections or implant, transdermal depot patch or vaginal ring). To be considered sterilised or infertile, females must have undergone surgical sterilisation (bilateral tubectomy, hysterectomy or bilateral ovariectomy) or be post-menopausal (defined as at least 12 months amenorrhoea and confirmed with follicle-stimulating hormone [FSH] test)

Exclusion Criteria:

1. Pregnancy or lactation
2. Positive results on the human immunodeficiency virus (HIV), hepatitis B and/or C tests
3. A history of clinically significant intestinal adhesions and/or chronic abdominal pain
4. Require chronic systemic narcotics for treatment of pain that exceeds an amount corresponding to 80 mg of morphine per day
5. History of cancer or clinically significant lymphoproliferative disease within ≤5 years, except for adequately treated basal cell skin cancer
6. History of gallstone within the past 3 years. Gallstone with subsequent cholecystectomy to resolve the issues is acceptable.
7. Inflammatory bowel disease patients (IBD) who have NOT been on a stable drug treatment regimen for at least the past 4 weeks
8. Evidence of active IBD in the past 12 weeks
9. Visible blood in the stool within the last 3 months
10. Decompensated heart failure (New York Heart Association [NYHA] class III-IV, see Appendix 12.2) and/or known coronary heart disease defined as unstable angina pectoris and/or myocardial infarction within the last 6 months prior to screening
11. Radiation enteritis, scleroderma or other condition of intestinal dysmotility, coeliac disease, refractory or tropical sprue
12. History of alcohol and/or drug abuse within the last 12 months
13. Inadequate hepatic function as defined by: bilirubin >upper limit of normal (ULN), alanine transaminase (ALT) or aspartate transaminase (AST) >2.0 × ULN; alkaline phosphatase (ALP) >2.5 × ULN; or international normalised ratio (INR) >1.5 × ULN
14. Inadequate renal function as defined by serum creatinine or blood urea nitrogen >2.5 x ULN
15. Unplanned hospitalisation of >24 hours duration within 1 month before the screening visit
16. Systemic corticosteroids, methotrexate, cyclosporine, tacrolimus, sirolimus, infliximab, or other biologic therapy/immune modifiers within 30 days of screening
17. Any use of growth hormone, glutamine or growth factors such as native GLP-2 or GLP-2 analogue within the last 3 months
18. Any use of antibiotics within the last 30 days
19. Participation in another clinical trial within the last 3 months and during this trial
20. Previously been treated in this trial
21. Loss of blood or donation of blood or plasma >500 mL within 3 months prior to screening
22. Patient not capable of understanding or not willing to adhere to the trial visit schedules and other protocol requirements
23. For any other reason judged not eligible by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day -28 to Day 26 plus 6 weeks
  Adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Assessment of intestinal insufficiency and gut absorption | Day -28 to day 26
  Changes in the wet weight (g) of faecal excretion
Assessment of intestinal insufficiency and gut absorption | Day -28 and day 26
  Changes from baseline in lean body mass by DEXA scan.
Assessment of intestinal insufficiency and gut absorption | Day -28 and day 26
  Changes from baseline in bone mineral content by DEXA scan.
Assessment of intestinal insufficiency and gut absorption | Day -28 and day 26
  Changes from baseline in fat mass by DEXA scan.
Assessment of intestinal insufficiency and gut absorption | Day -28 to day 26 plus 6 weeks
  Measure of body weight (kg)
Assessment of intestinal insufficiency and gut absorption | Baseline (Day -6) to end of treatment (Day 26)
  Measurement of urinary output (ml)
Assessment of intestinal insufficiency and gut absorption | Baseline (Day -6) to end of treatment (Day 26)
  Measurement of urinary electrolytes (sodium, potassium, calcium, magnesium) (mmol/d)
Assessment of gut regeneration | Baseline (Day -7) to end of treatment period (Day 26) plus 6 weeks
  Measurements of the plasma Citrulline (ng/ml)
Maximum observed plasma concentration (Cmax) | Day 1 to end of treatment period (Day 26)
  Cmax (ng/ml)
Cumulative area under the plasma concentration (AUC) of FE 203799 from time 0 to 168 | Day 1 to end of treatment period (Day 26)
  AUC0-168 (ng*hr/ml)
Terminal elimination half-life (T1/2) of FE 203799 | Day 1 to end of treatment period (Day 26)
  T1/2 (h)
Apparent total body clearance (CL) of FE 203799 from plasma | Day 1 to end of treatment period (Day 26)
  CL (ml/hr)
Apparent volume of distribution (Vd) of FE 203799 during terminal phase | Day 1 to end of treatment period (Day 26)
  Vd (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No